CLINICAL TRIAL: NCT00690053
Title: Non-Invasive Imaging of [18F]HX4 With Positron-Emission-Tomography (PAT): A Phase I Study
Brief Title: Non-Invasive Imaging of [18F]HX4 With Positron-Emission-Tomography (PET)
Acronym: HX-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: dr. D.K.M. De Ruysscher, Maastro Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 08-3-040
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-02

CONDITIONS: Cancer
Keywords: Toxicity; PET; HX-4; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Injection of HX-4

INTERVENTIONS:
Procedure: Injection of HX-4 — In step 1: 1 injection of HX-4 (max.6mCi (222MBq)) In step 2: 1 injection of HX-4 (max.12mCi 444MBq)

SUMMARY:
Non invasive imaging of hypoxia with the aid of PET-scans could help to select the patients having a hypoxic tumour who could be treated with specific anti-hypoxic treatments such as bio-reductive drugs or hypoxic radio-sensitizers. Several 2-nitroimidazoles to which the compound to be tested, HX-4, belongs, labelled with Fluor-18 have already been used in patients. However, bad image quality and unpredictable kinetics limit their use. In extensive pre-clinical models, the combination of HX-4 labelled with Fluor-18 is a promising non-toxic new probe to determine hypoxia.

DETAILED DESCRIPTION:
To determine the toxicity of the hypoxia PET-tracer [18F]-HX4 in cancer patients in two dose-steps:

* Step 1 (3-6 patients): a single dose of maximum 6 mCi (222 MBq) dose of [18F]HX4 (which contains a maximum of 15 μg HX-4) via a bolus IV injection.
* Step 2 (3-6 patients): a single dose of maximum 12 mCi (444 MBq) dose of [18F]HX4 (which contains a maximum of 27 μg HX-4) via a bolus IV injection.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed solid tumour, primary or secondary stage IV and/ or tumours with no curative treatment options.
* Normal white blood cell count and neutrophils
* Normal platelet count
* No anaemia requiring blood transfusion or erythropoietin
* Adequate hepatic function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution).
* Calculated Creatinin clearance at least 60 ml/min
* No administration of Fluor-18 in the previous 24 hours
* Capable of complying with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Toxicity (CTCAE 3.0) | 9 months

SECONDARY OUTCOMES:
Image Quality at different time points (Tumour-to-Background Ratio determined by PET-CT scan) | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht Radiation Oncology (MAASTRO clinic), Maastricht, Netherlands